CLINICAL TRIAL: NCT04541667
Title: Is End Tidal CO2 Level Elevation During Upper Endoscopy With CO2 Gas Insufflation Physiologically Significant
Acronym: ETCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Children's Hospital and Medical Center, Omaha, Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0632-19-FB
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Endoscopy
Keywords: upper endoscopy; endoscope; abdominal discomfort; insufflation; carbon dioxide
MeSH Terms: interventions — Air; Gases; Carbon Dioxide

STUDY DESIGN:
Intervention Model Description: Eligible study participants will be randomized 1:1 into two study arms; one receiving air and the other receiving carbon dioxide for luminal inflation.
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded, prospective, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Air for luminal inflation (Active Comparator): Patients randomized into this arm will have luminal inflation using air.
  Interventions: Other: Air
- Carbon Dioxide for luminal inflation (Active Comparator): Patients randomized into this arm will have luminal inflation using carbon dioxide.
  Interventions: Other: Carbon Dioxide

INTERVENTIONS:
Other: Air — Air will be used for luminal inflation.
  Other Names: Gas
  Arms: Air for luminal inflation
Other: Carbon Dioxide — Carbon dioxide will be used for luminal inflation.
  Other Names: Gas
  Arms: Carbon Dioxide for luminal inflation

SUMMARY:
During the course of an endoscopic procedure, air has historically been used to inflate the lumen to provide adequate visualization and allow for the endoscope to advance as necessary. In many adult centers, carbon dioxide is used for insufflation for all procedures. Many pediatric centers have started using carbon dioxide for insufflation during endoscopy based on the adult studies. Few pediatric studies have been done. This study is designed to test whether carbon dioxide is associated with any negative, post-procedural, outcomes in pediatric patients.

DETAILED DESCRIPTION:
Luminal inflation is essential for adequate visualization and endoscope advancement during endoscopy. Although air has previously been the standard gas used, CO2 is increasing preferred in adult endoscopy centers, due to reports of decreased post-procedural abdominal discomfort compared to air. Few published studies in children demonstrated decreased abdominal discomfort with use of CO2, but safety concerns for its use in pediatric endoscopy remain.

This is a Double-blinded, prospective, randomized study of all pediatric patients undergoing procedures involving upper endoscopy in the Childrens Hospital & Medical Center. Randomization will be for patients undergoing upper endoscopy related procedures. Patients will be randomized 1:1 for air or CO2. Vital signs will be recorded before the procedure, throughout the procedure and after the procedure until fully awake. While in the procedure room, end-tidal CO2 level will be continuously recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 months to 19 years old and
* Undergoing upper endoscopy at Children's Hospital & Medical Center in Omaha, NE and
* Parents or legal guardians consent to the study

Exclusion Criteria:

* Patients and legal guardians who decline participation in the study
* Patients with chronic respiratory disease (defined as severe asthma, bronchopulmonary dysplasia and cystic fibrosis-related pulmonary disease)
* Patients with cyanotic heart disease
* Patients with an ASA status of ≥ 3.
* Patients who are wards of the state or in foster care
* Prisoners
* Patients undergoing colonoscopy only procedures or procedures not related to upper endoscopy

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chinenye R Dike, MD, Principal Investigator — Children's Hospital & Medical Center / University of Nebraska Medical Center
Locations (1):
- Children's Hospital & Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steppan J, Hogue CW Jr. Cerebral and tissue oximetry. Best Pract Res Clin Anaesthesiol. 2014 Dec;28(4):429-39. doi: 10.1016/j.bpa.2014.09.002. Epub 2014 Sep 28. PMID 25480772
- [Background] ASGE Technology Committee; Lo SK, Fujii-Lau LL, Enestvedt BK, Hwang JH, Konda V, Manfredi MA, Maple JT, Murad FM, Pannala R, Woods KL, Banerjee S. The use of carbon dioxide in gastrointestinal endoscopy. Gastrointest Endosc. 2016 May;83(5):857-65. doi: 10.1016/j.gie.2016.01.046. Epub 2016 Mar 3. No abstract available. PMID 26946413
- [Background] Chen SW, Hui CK, Chang JJ, Lee TS, Chan SC, Chien CH, Hu CC, Lin CL, Chen LW, Liu CJ, Yen CL, Hsieh PJ, Liu CK, Su CS, Yu CY, Chien RN. Carbon dioxide insufflation during colonoscopy can significantly decrease post-interventional abdominal discomfort in deeply sedated patients: A prospective, randomized, double-blinded, controlled trial. J Gastroenterol Hepatol. 2016 Apr;31(4):808-13. doi: 10.1111/jgh.13181. PMID 26421801
- [Background] Liu X, Liu D, Li J, Ou D, Zhou Z. [Safety and efficacy of carbon dioxide insufflation during colonoscopy]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2009 Aug;34(8):825-9. Chinese. PMID 19734597
- [Background] Lynch I, Hayes A, Buffum MD, Conners EE. Insufflation using carbon dioxide versus room air during colonoscopy: comparison of patient comfort, recovery time, and nursing resources. Gastroenterol Nurs. 2015 May-Jun;38(3):211-7. doi: 10.1097/SGA.0000000000000109. PMID 25946475
- [Background] Memon MA, Memon B, Yunus RM, Khan S. Carbon Dioxide Versus Air Insufflation for Elective Colonoscopy: A Meta-Analysis and Systematic Review of Randomized Controlled Trials. Surg Laparosc Endosc Percutan Tech. 2016 Apr;26(2):102-16. doi: 10.1097/SLE.0000000000000243. PMID 26841319
- [Background] Riss S, Akan B, Mikola B, Rieder E, Karner-Hanusch J, Dirlea D, Mittlbock M, Weiser FA. CO2 insufflation during colonoscopy decreases post-interventional pain in deeply sedated patients: a randomized controlled trial. Wien Klin Wochenschr. 2009;121(13-14):464-8. doi: 10.1007/s00508-009-1202-y. PMID 19657610
- [Background] Sajid MS, Caswell J, Bhatti MI, Sains P, Baig MK, Miles WF. Carbon dioxide insufflation vs conventional air insufflation for colonoscopy: a systematic review and meta-analysis of published randomized controlled trials. Colorectal Dis. 2015 Feb;17(2):111-23. doi: 10.1111/codi.12837. PMID 25393051
- [Background] Singh R, Neo EN, Nordeen N, Shanmuganathan G, Ashby A, Drummond S, Nind G, Murphy E, Luck A, Tucker G, Tam W. Carbon dioxide insufflation during colonoscopy in deeply sedated patients. World J Gastroenterol. 2012 Jul 7;18(25):3250-3. doi: 10.3748/wjg.v18.i25.3250. PMID 22783048
- [Background] Homan M, Mahkovic D, Orel R, Mamula P. Randomized, double-blind trial of CO2 versus air insufflation in children undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):993-7. doi: 10.1016/j.gie.2015.08.073. Epub 2015 Sep 10. PMID 26363332
- [Background] Kresz A, Mayer B, Zernickel M, Posovszky C. Carbon dioxide versus room air for colonoscopy in deeply sedated pediatric patients: a randomized controlled trial. Endosc Int Open. 2019 Feb;7(2):E290-E297. doi: 10.1055/a-0806-7060. Epub 2019 Jan 30. PMID 30705964
- [Background] Thornhill C, Navarro F, Alabd Alrazzak B, Hashmi SS, DebRoy AN, Rhoads JM, Imseis E. Insufflation With Carbon Dioxide During Pediatric Colonoscopy for Control of Postprocedure Pain. J Clin Gastroenterol. 2018 Sep;52(8):715-720. doi: 10.1097/MCG.0000000000000910. PMID 29210902
- [Background] Eastwood GM, Tanaka A, Bellomo R. Cerebral oxygenation in mechanically ventilated early cardiac arrest survivors: The impact of hypercapnia. Resuscitation. 2016 May;102:11-6. doi: 10.1016/j.resuscitation.2016.02.009. Epub 2016 Feb 21. PMID 26903288
- [Background] Erdogan S, Oto A, Bosnak M. Reliability of cerebral oximeter in non-invasive diagnosis and follow-up of hypercapnia. Turk J Pediatr. 2016;58(4):389-394. doi: 10.24953/turkjped.2016.04.007. PMID 28276211
- [Derived] Dike CR, Huang Pacheco A, Lyden E, Freestone D, Choudhry O, Bishop WP, Shukry M. Elevations in End-Tidal CO 2 With CO 2 Use During Pediatric Endoscopy With Airway Protection: Is This Physiologically Significant? J Pediatr Gastroenterol Nutr. 2023 May 1;76(5):660-666. doi: 10.1097/MPG.0000000000003748. Epub 2023 Feb 22. PMID 36821847

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant who consented withdrew consent prior to randomization. Therefore, this patient did not undergo randomization
Units Other Than Participants: Procedures
Period: Overall Study
Arm/Group | Air for Luminal Inflation | Carbon Dioxide for Luminal Inflation
Started | 98; 98 Procedures | 102; 102 Procedures
Completed | 98; 98 Procedures | 102; 102 Procedures
Not Completed | 0; 0 Procedures | 0; 0 Procedures

BASELINE CHARACTERISTICS:
Population: Population was mostly female, Caucasians and older children
Units Other Than Participants: Procedures
Groups:
- Total: Total of all reporting groups
Arm/Group | Air for Luminal Inflation | Carbon Dioxide for Luminal Inflation | Total
Number analyzed (Participants) | 98 | 102 | 200
Number analyzed (Procedures) | 98 | 102 | 200
Age, Continuous [Median (Full Range); unit: years] | 12 [0 to 19] | 12 [1 to 19] | 12 [0 to 19]
Sex: Female, Male [Count of Units; unit: Procedures]
  Female | 58 | 56 | 114
  Male | 40 | 46 | 86
Ethnicity (NIH/OMB) [Count of Units; unit: Procedures]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 92 | 96 | 188
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: Procedures]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 84 | 84 | 168
  More than one race | 6 | 10 | 16
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 98 | 102 | 200
BMI z score [Median (Full Range); unit: units on a scale] — This represents a scale of mean with standard deviations from the mean. For example z score of 0 is at mean. Z score of + 1 represents 1 SD from the mean and z score of -1 represents 1 SD below the mean. Z scores of > or = -1 represent malnutrition. Z
  units on a scale | 0.23 [-3.86 to 2.94] | 0.61 [-2.90 to 2.72] | 0.23 [-3.86 to 2.94]

OUTCOME MEASURES:

1. Primary Outcome: Number of Procedures With Elevated End-tidal CO2 Levels
Description: Compare the peak end-tidal CO2 levels (>/= 60 mmHg) observed during endoscopy in children managed with endotracheal intubation or laryngeal mask airway using CO2 versus air
Time Frame: Measured from time of procedure start to time of procedure conclusion this lasts usually from 1-2.5 hours.
Population: Participants in this groups refers to procedures. Procedure count was used for analysis and not participant count
Measure: Count of Units; unit: Procedures
Units Other Than Participants: Procedures
Groups:
- Air for Luminal Inflation: Procedures randomized into this arm will have luminal inflation using air.
  Air: Air will be used for luminal inflation.
- Carbon Dioxide for Luminal Inflation: Procedures randomized into this arm will have luminal inflation using carbon dioxide.
  Carbon Dioxide: Carbon dioxide will be used for luminal inflation.
Arm/Group | Air for Luminal Inflation | Carbon Dioxide for Luminal Inflation
Number analyzed (Participants) | 98 | 102
Number analyzed (Procedures) | 98 | 102
Procedures | 8 | 21

2. Secondary Outcome: Number of Participants Reporting Abdominal Pain
Description: Pain rating scales using FLACC and VAS will be used to assess self reported pain before and after the procedure
Time Frame: This will be assessed before and after the procedure
Population: Participant procedures randomized into air or CO2 for endoscopic insufflation. Participants reporting abdominal pain after procedure. Higher numbers are worse
Measure: Number; unit: participants
Arm/Group | Air for Luminal Inflation | Carbon Dioxide for Luminal Inflation
Number analyzed (Participants) | 97 | 102
participants | 14 | 15

ADVERSE EVENTS:
Time Frame: Procedure duration which lasts between 1-2.5 hours
Description: Procedure related adverse events such as bleeding and perforation Anesthesia related adverse events such as hypotension, hypertension, tachypnea
Arm/Group | Air for Luminal Inflation | Carbon Dioxide for Luminal Inflation
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/102
Other Adverse Events (participants affected / at risk) | 5/98 | 5/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Air for Luminal Inflation (N=98) | Carbon Dioxide for Luminal Inflation (N=102)
Hypotension (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 2 | 2
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT04541667/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04541667/ICF_001.pdf